CLINICAL TRIAL: NCT02955953
Title: Bioequivalence Study Comparing the Pharmacokinetics and Glucodynamics of LY2963016 U-200 Formulation With LY2963016 U-100 Formulation in Healthy Subjects
Brief Title: A Study Comparing Two Formulations of Insulin Glargine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16249; I4L-MC-ABEV (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-11-03; First posted 2016-11-04 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — LY2963016 insulin glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2963016 U-200 Formulation (Test) (Experimental): LY2963016 test formulation administered as a subcutaneous (SC) injection in one of two or two of four study periods.
  Interventions: Drug: LY2963016
- LY2963016 U-100 Formulation (Reference) (Experimental): LY2963016 reference formulation administered as a SC injection in one of two or two of four study periods.
  Interventions: Drug: LY2963016

INTERVENTIONS:
Drug: LY2963016 — Administered SC

SUMMARY:
The study will aim to evaluate the following:

* Whether there are any differences in the way the body handles LY2963016 U-200 and LY2963016 U-100.
* How well-tolerated LY2963016 U-200 is compared with LY2963016 U-100.
* How LY2963016 U-200 affects the level of blood sugar in the body compared with LY2963016 U-100.

The study will last up to 17 weeks for each participant, including initial screening and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m²)
* Have a fasting plasma glucose less than (<) 6.0 millimoles per liter (mmol/L) (108 milligram per deciliter [mg/dL])
* Have venous access sufficient to allow for blood sampling and clamp procedures per protocol

Exclusion Criteria:

* Have known allergies to the study drug, or any components of the formulation
* Have donated or had a blood loss of 450 milliliter (mL) within 3 months prior to study enrollment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of LY2963016 U-200 Formulation and LY2963016 U-100 Formulation | One hour before dosing up to 48 hours following administration of study drug
Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) of LY2963016 U-200 Formulation and LY2963016 U-100 Formulation | One hour before dosing up to 48 hours following administration of study drug

SECONDARY OUTCOMES:
Pharmacodynamics: Total Amount of Glucose Infused (Gtot) of LY2963016 U-200 and LY2963016 U-100 | One hour before dosing up to about 30 hours post clamp procedure
Pharmacodynamics: Maximum Glucose Infusion Rate (Rmax) of LY2963016 U-200 and LY2963016 U-100 | One hour before dosing up to about 30 hours post clamp procedure

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore